CLINICAL TRIAL: NCT07299071
Title: Randomized Controlled Trial Evaluating the Efficacy of CAD in Screening Colonoscopy to Reduce the Risk of Advanced Adenoma at 3 Years.
Brief Title: Efficacy of CAD in Screening Colonoscopy to Reduce the Risk of Advanced Adenoma at 3 Years.
Acronym: IA-COLO 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CHUBX 2024/48
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Colonoscopy; Colorectal Neoplasms; Intestinal Polyps
Keywords: colonoscopy; colorectal neoplasms; computer aided diagnosis
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Polyps

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard colonoscopy (Placebo Comparator): Patients will be enrolled after a pre-colonoscopy consultation and risk-assessment for colorectal cancer. The screening colonoscopy will be performed by an investigator. Patients will be randomized in the endoscopy room after confirmed cecal intubation and quality of bowel preparation. Patient has standard colonoscopy
  Interventions: Procedure: Standard colonoscopy
- Colonoscopy with CADe (Active Comparator): Patients will be enrolled after a pre-colonoscopy consultation and risk-assessment for colorectal cancer. The screening colonoscopy will be performed by an investigator. Patients will be randomized in the endoscopy room after confirmed cecal intubation and quality of bowel preparation. Patient has colonoscopy with CADe (CAD EYE or GENIUS)
  Interventions: Procedure: Colonoscopy CADe

INTERVENTIONS:
Procedure: Standard colonoscopy — Colonoscopy standard (without CADe)
  Arms: Standard colonoscopy
Procedure: Colonoscopy CADe — colonoscopy with CADe
  Arms: Colonoscopy with CADe

SUMMARY:
The occurrence of interval cancers after colonoscopy raises the possibility of missed lesions. High- performance computer aided diagnosis (CAD) systems have been specially designed for the detection of colorectal lesions (CAD for detection is named CADe). The use of CADe improves adenoma detection in screening colonoscopy. The potential of CADe system in reducing the rate of progression to advanced polyps or interval cancer between two colonoscopies remains still uncertain.

DETAILED DESCRIPTION:
Patients will be enrolled after a pre-colonoscopy consultation and risk-assessment for colorectal cancer. The screening colonoscopy will be performed by an investigator. Patients will be randomized in the endoscopy room after confirmed cecal intubation and quality of bowel preparation. Randomization into two groups: standard colonoscopy vs. colonoscopy with CADe (CAD EYE or GENIUS) (1:1). A follow-up consultation will be scheduled one-month postcolonoscopy for delivery of histological results and then at 3 years in order to organize the next colonoscopy. As part of the study, a new control colonoscopy will be scheduled for patients with high risk of CRC at 3 years. The 3-year control colonoscopy will be performed with the CAD system for all patients. The colonoscopy will be performed by another investigator who does not know the results nor the type of the first colonoscopy (evaluator blinded). In the low-risk group, we will collect follow-up data as part of routine care, including the results of colonoscopies performed outside of the protocol

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with indication for colonoscopy as part of a screening program, after a positive immunological (FIT) test, and/or for personal or family history of colorectal cancer and/or personal history of colonic adenomas,
* Written informed consent signed
* Patients covered by a health-care insurance.

Exclusion Criteria:

* Failed complete colonoscopy, defined by the absence of cecal intubation and/or the absence of terminal ileum cauterization
* Inadequate bowel preparation (Boston bowel preparation score < 6, and/or least at one part of colon with score ≤ 1)
* An infiltrative tumor was diagnosed during colonoscope insertion time, not accessible to endoscopic resection and likely to require surgical management (a procedure where part of the colon may need to be removed).
* Patient under guardianship or protection
* Pregnant women
* Not fluent in French or illiterate
* Personal history of inflammatory bowel disease
* Personal history of genetic predisposition of CRC
* Personal history of colonic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Advanced adenoma | 36 months
  The proportion of patients presenting at least one advanced adenoma detected after a 3-year follow-up period. An advanced adenoma is defined as an adenoma or sessile serrate adenoma (SSL) larger than 1cm (size confirmed by the CAD system and/or size estimation by snare), and/or with high-grade dysplasia or neoplasia (confirmed by histological analysis).

SECONDARY OUTCOMES:
Number of adenoma | 36 months
  Average number of adenoma or SSL (confirmed by histological analysis) detected in each patient during screening colonoscopy after a 3-year follow-up period
Estimation of the sensitivity of CADx | Day0, 36 months
  Estimated sensitivity of CADx (CAD for characterization is named CADx) for the diagnosis and evaluation of colonic polyp's malignancy, with histologic analysis in each center as a reference diagnosis.
Estimation of the specificity of CADx | DAY 0, 36 months
  Estimated specificity of CADx (CAD for characterization is named CADx) for the diagnosis and evaluation of colonic polyp's malignancy, with histologic analysis in each center as a reference diagnosis.
Cost of CADe and classical colonoscopy | Day 0, 36 months
  The cost of CADe and classical colonoscopy will be estimated using a bottom-up micro costing approach

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CH de la Côte Basque, Bayonne
  - CHU Brest la Cavale Blanche, Brest
  - Clinique Paris Bercy, Charenton-le-Pont
  - CHU de Limoges, Limoges
  - Institut Paoli Calmettes, Marseille
  - Clinique Jules Verne, Nantes
  - CHU Nîmes, Nîmes
  - APHP - Hôpital Saint Antoine, Paris
  - Aphp-Hegp, Paris
  - CHU Bordeaux - Hôpital Haut Lévêque, Pessac
  - CHU de Rennes, Rennes
  - Clinique Pasteur, Toulouse
  - CHRU de Nancy - Hôpital Brabois Adultes, Vandœuvre-lès-Nancy